CLINICAL TRIAL: NCT00461916
Title: Half-Dose Depot Triptorelin Versus Reduced-Dose Daily Buserelin in a Long Protocol of Controlled Ovarian Stimulation for ICSI/ET
Brief Title: Half-Dose Depot Triptorelin Versus Reduced-Dose Daily Buserelin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5152
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Infertility
Keywords: half-dose depot triptorelin; reduced-dose daily buserelin; controlled ovarian stimulation; long protocol; ICSI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Half-Dose Depot Triptorelin
Drug: Reduced-Dose Daily Buserelin

SUMMARY:
The purpose of this study is to determine whether half-dose depot triptorelin are as effective as reduced-dose daily buserelin in the controlled ovarian stimulation for intracytoplasmic sperm injection and embryo transfer

DETAILED DESCRIPTION:
Significant doubts remain about which type of GnRH agonists [GnRHa] administration to be used in controlled ovarian stimulation [COS] cycles. The use of a single-dose depot long-acting GnRHa instead of a daily low dose preparation would be more comfortable for patients, however, inducing a profound pituitary desensitization, it increases the number of gonadotropin ampoules and the duration of the COS cycle without improving pregnancy rates or other clinical outcomes. Thus, some authors recommend a reduction of both dose and/or duration of GnRHa administration. Halving the dose of depot triptorelin, for instance, has been studied against its full dose administration since 1992 with rather similar clinical outcomes. Half-dose depot leuprolide acetate has also resulted in comparable clinical outcomes with standard daily injections in long GnRHa protocol. Reducing the daily doses of short acting GnRHa has been advocated to demonstrate equivalent results to standard doses. To our knowledge, however, the reduced daily doses have not been evaluated against half dose depot forms in long GnRHa protocols.

Thus, we originally compared a half-dose depot triptorelin with reduced daily doses of short-acting buserelin in a long protocol for intracytoplasmic sperm injection and embryo transfer [ICSI/ET] cycles.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for ICSI/ET
* 35 years old or younger
* Serum FSH less than 10 IU/l on day three of the previous menstrual cycle
* No more than two previous IVF/ICSI attempts
* No planned percutaneous epididymal sperm aspiration [PESA]
* No planned testicular sperm extraction [TESE]
* No known history or risk of severe hyperstimulation
* No evidence of hydrosalpinx
* No major systemic disease
* No uterine abnormality
* No previous ovarian surgery

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182
Dates: Start 2005-05; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of retrieved oocytes

SECONDARY OUTCOMES:
Number of days of gonadotropin stimulation
Number of hMG ampoules
Number of follicles at hCG administration
Quality of oocytes
Quality of embryos
Poor response rate
Oocyte fertilization rate
Ineffective intervention rate
Clinical pregnancy rate
Implantation rate
Biochemical pregnancy rate
Multiple pregnancy rate
Miscarriage rate
Ectopic pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Leili Safdarian, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Dr. Shariati Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Safdarian L, Mohammadi FS, Alleyassin A, Aghahosseini M, Meysamie A, Rahimi E. Clinical outcome with half-dose depot triptorelin is the same as reduced-dose daily buserelin in a long protocol of controlled ovarian stimulation for ICSI/embryo transfer: a randomized double-blind clinical trial (NCT00461916). Hum Reprod. 2007 Sep;22(9):2449-54. doi: 10.1093/humrep/dem223. Epub 2007 Jul 17. PMID 17635844